CLINICAL TRIAL: NCT02823327
Title: Clinical and Genomic Factors for Prognosis of AIDS Primary Effusion Lymphoma
Status: Terminated | Type: Observational
Why Stopped: Poor accrual
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, San Diego (Other); University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: AMC-S004; NCI-2015-00794 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-S004 (Other: National Cancer Institute); AMC #S004 (Other: AMC); S004 (Other: AMC); AMC-S004 (Other: AIDS Malignancy Consortium); AMC-S004 (Other: CTEP); U01CA121947 (NIH)
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: AIDS-Related Primary Effusion Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissues slides for verification of pathological diagnosis of primary effusion lymphoma.
  Paraffin embedded tissues or cytology block or frozen tissue specimen for genomic analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chart review, RNA sequencing, microarray: Laboratory Biomarker Analysis. Medical chart review is performed and patient information is collected regarding human immunodeficiency virus HIV/AIDS medical history, staging of AIDS related malignancy, and type of treatment. Previously collected tissue samples are analyzed via RNA sequencing and microarray.
  Interventions: Genetic: Laboratory Biomarker Analysis; Other: Medical Chart Review

INTERVENTIONS:
Genetic: Laboratory Biomarker Analysis — Correlative studies
Other: Medical Chart Review — Medical chart review is performed
  Other Names: Chart Review

SUMMARY:
This research trial studies clinical factors and gene expression analysis for prognosis in tissue samples from patients with acquired immune deficiency syndrome (AIDS)-related primary effusion lymphoma. Gathering health information over time and studying samples of tissue from patients in the laboratory may help doctors learn about the prognosis of patients with AIDS-related primary effusion lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify baseline clinical characteristics and treatment strategies in patients with AIDS-associated primary effusion lymphoma (PEL) that correlate with long-term survival (>= 2 years). (Primary clinical objective) II. Identify differentially expressed genes in PEL that are associated with long-term survival (>= 2 years). (Primary genomic objective)

OUTLINE:

Medical chart review is performed and patient information is collected regarding human immunodeficiency virus human immunodeficiency virus (HIV)/AIDS medical history, staging of AIDS related malignancy, and type of treatment. Previously collected tissue samples are analyzed via ribonucleic acid (RNA) sequencing and microarray.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary effusion lymphoma (HIV seropositive or negative) on or after January 1, 1998 on whom survival status at 2 years post PEL diagnosis is available
* Participants may be enrolled to either or both the clinical or genomic portions of the study
* The minimum data required to be able to include a subject for analysis of clinical prognostic factors are:

  * HIV status, and for HIV subjects include cluster of differentiation (CD)4 count, HIV viral load closest to time of diagnosis
  * Age at PEL diagnosis
  * Gender
  * Stage at diagnosis
  * Treatment of PEL
  * Response to treatment
  * Survival status at 2 years
  * Pathology slides (or paraffin block) for central review
* The minimum data required to be able to include a subject for analysis of genomic prognostic factors are:

  * Availability of a pathologic specimen of PEL that will be submitted for genomic analysis
  * Survival status at 2 years

Exclusion Criteria:

* Patients who do not fulfill the criteria as listed above are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with primary effusion lymphoma (HIV seropositive or negative) on or after January 1, 1998 and on whom survival status at 2 years post diagnosis is available.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Reid, Principal Investigator — AIDS Malignancy Consortium
Locations (6):
- United States (6):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA CARE Center, Los Angeles, California
  - University of Miami, Miami, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chart Review, RNA Sequencing, Microarray
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chart Review, RNA Sequencing, Microarray
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 3
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54.7 [48 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 14
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 25
HIV status [Count of Participants; unit: Participants]
  HIV positive | 24
  HIV negative | 1
HAART receipt at any time prior to PEL diagnosis [Count of Participants; unit: Participants]
  Yes | 16
  No | 8
  Unknown | 1
HARRT at the time of PEL diagnosis [Count of Participants; unit: Participants]
  Yes | 18
  No | 6
  Unknown | 1
History of Kaposi Sarcoma (KS) [Count of Participants; unit: Participants]
  Yes | 11
  No | 13
  Unknown | 1
Prior treatment for KS [Count of Participants; unit: Participants] — Population: Among 25 participants, there were 11 participants received KS treatment.
  Participants
    number analyzed (Participants) | 11
    Yes | 5
    No | 6
KS treatment within 1 month prior to PEL diagnosis [Count of Participants; unit: Participants] — Population: Among 11 participants received KS treatment, there were 5 participants received prior treatment.
  Participants
    number analyzed (Participants) | 5
    Yes | 2
    No | 3
History of MCD [Count of Participants; unit: Participants]
  Yes | 5
  No | 19
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Differential Gene Expression Profile by RNA-Seq or GeneChip Assays
Description: The resultant data will be a subset of the whole analysis population due to RNAseq data availability. It will be assessed for quality, normalized, and then analyzed for differential gene expression. The Nanostring software nSolver will be used to do quality control, background subtraction, normalization, and analysis of the differential expression for RNA-sequencing data. Lastly, bioinformatic analysis approaches will be used to help make sense of possible biological links between the genes found to be differentially expressed between the sample groups that may be of prognostic significance. 19 Genes with p-value less than 0.05 were reported by the level of gene expression.
Time Frame: baseline
Population: RNAseq data were available from 20 participants among 25 participants.
Measure: Number; unit: Number of overexpressed genes
Groups:
- Survival Less Than 2 Years With Available RNAseq Data: 7 participants had RNAseq data among 8 participants with survival less than 2 years.
- Survival More Than or Equal to 2 Years With Available RNAseq Data: 13 participants had RNAseq data among 17 participants with survival more than or equal to 2 years.
Arm/Group | Survival Less Than 2 Years With Available RNAseq Data | Survival More Than or Equal to 2 Years With Available RNAseq Data
Number analyzed (Participants) | 7 | 13
Number of overexpressed genes | 4 | 15

2. Primary Outcome: Response Rates
Description: The number of participants for this outcome measure is 25 participants with baseline characteristics and response evaluation. Since this was a retrospective study, response criteria were not defined. Response determinations as recorded in the medical record by the treating physician were abstracted on each participant for data analysis. Response rates will be reported with 95% confidence intervals (binomial distribution). Descriptive statistics will be used to summarize baseline clinical, histological, and viral characteristics.
Time Frame: Up to 1 year
Population: Response rates for the first line of therapy were estimated by survival status.
Measure: Count of Participants; unit: Participants
Groups:
- Survival Less Than 2 Years: 8 participants with survival less than 2 years
- Survival More Than or Equal to 2 Years: 17 participants with survival more than or equal to 2 years
Arm/Group | Survival Less Than 2 Years | Survival More Than or Equal to 2 Years
Number analyzed (Participants) | 8 | 17
Participants
  Complete response | 1 | 13
  Partial response | 2 | 2
  Stable disease | 2 | 2
  Progression | 3 | 3

3. Primary Outcome: Survival Status at 2 Years
Description: Survival duration will be determined using the elapsed time between the date of PEL diagnosis and the last follow-up date or the date of death.
Time Frame: At 2 years post diagnosis
Population: There are 8 participants with survival less than 2 years and 17 participants with survival more than or equal to 2 years.
Measure: Number; unit: participants
Groups:
- Survival Less Than 2 Years: Survival status at 2 years was determined using medical chart review for 25 participants. There were 8 participants with survival less than 2 years.
- Survival More Than or Equal to 2 Years: Survival status at 2 years was determined using medical chart review for 25 participants. There were 17 participants with survival more than or equal to 2 years.
Arm/Group | Survival Less Than 2 Years | Survival More Than or Equal to 2 Years
Number analyzed (Participants) | 8 | 17
participants
  Hispanic | 2 | 5
  Non-Hispanic | 6 | 12
  White | 5 | 9
  Non-White | 3 | 8
  EPOCH treatment | 4 | 13
  Non-EPOCH treatment | 4 | 4
  Stage I-III | 2 | 6
  Stage IV | 6 | 11

ADVERSE EVENTS:
Time Frame: This study is a retrospective, chart-review study. The time frame for evaluating adverse event is not applicable.
Description: This study is a retrospective, chart-review study. Death and Adverse Events were not assessed. The adverse event report is not relevant. Since this is not an interventional study, the adverse event report is not relevant.
Arm/Group | Chart Review, RNA Sequencing, Microarray
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT02823327/Prot_SAP_000.pdf